CLINICAL TRIAL: NCT05383105
Title: Virtual Bronchoscopic Navigation to Increase Diagnostic Yield in Patients With Pulmonary Nodules
Acronym: NAVIGATOR
Status: Recruiting | Type: Observational
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Principal Investigator, Dirk-Jan Slebos, Md PhD, University Medical Center Groningen
Other Study IDs: 202100352
Record Dates: First submitted 2022-05-16; First posted 2022-05-19 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: Pulmonary Nodules, Solitary
MeSH Terms: conditions — Solitary Pulmonary Nodule

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Virtual bronchoscopic navigation — Virtual bronchoscopy navigation (VBN) calculates the access to a solitary pulmonary nodule via a trans-parenchymal route. In contrast to the gold Standard transthoracic approach, with this technique also very small lesions (7 mm diameter), and lesions which cannot be reached via the transthoracic route - located in the inner two thirds of the lung - can be approached.
  Other Names: Archimedes

SUMMARY:
Background Transthoracic computed tomography (CT)-guided procedures are the current gold Standard for obtaining diagnostic biopsies of solitary pulmonary nodules (SPN) in the peripheral lung. Novel endobronchial techniques, such as electromagnetic navigation bronchoscopy (ENB) or Virtual bronchoscopic navigation (VBN) are considered safer to approach SPNs.

The newest technique combines VBN with calculating the access to a SPN via a transparenchymal route. In contrast to the gold Standard transthoracic approach, also small lesions, and lesions which cannot be reached transthoracicaliy, located in the innertwo thirdsof the lung can be approached.

Main research question To assess diagnostic yield of the novel Standard of care 'Virtual bronchoscopy navigation" procedure.

Design (including population, confounders/outcomes) A single centre, prospective, observational study of patients undergoing the novel Standard of care Virtual bronchoscopy navigation procedure to assess a pulmonary nodule. Clinical data of at least 100 consecutive patients will be collected.

DETAILED DESCRIPTION:
Background Transthoracic computed tomography (CT)-guided procedures are the current gold Standard for obtaining diagnostic biopsies of solitary pulmonary nodules (SPN) in the peripheral lung. Despite its accuracy and diagnostic yield, this technique is associated with an increased risk of complications, Pneumothorax and severe bleeding are the most frequent complications occurring in up to 27% of cases each.

Novel endobronchial techniques, such as electromagnetic navigation bronchoscopy (ENB) or Virtual bronchoscopic navigation (VBN) are considered safer to approach SPNs. The overall rate of pneumothorax after ENB is 4.3%, and bleeding occurs in only 2.8% of cases. The combination of techniques led to an overall increase of the diagnostic yield.

The newest technique combines VBN with calculating the access to a SPN via a transparenchymal route. In contrast to the gold Standard transthoracic approach, also small lesions, and lesions which cannot be reached transthoracicaliy, located in the innertwo thirdsof the lung can be approached. Detailed clinical data, like the correlation of the diagnostic yield to the specific location of the pulmonary nodule, however, is lacking. In view of the expected lung cancer screening program leading to increasing numbers of especially small pulmonary nodules, this data, however, is considered useful to help to select patients forthe right diagnostic procedure.

Main research question To assess diagnostic yield of the novel Standard of care 'Virtual bronchoscopy navigation" procedure.

Design (including population, confounders/outcomes) A single centre, prospective, observational study of patients undergoing the novel Standard of care Virtual bronchoscopy navigation procedure to assess a pulmonary nodule. Clinical data of at least 100 consecutive patients will be collected.

Expected results With the VBN procedure a histologie diagnosis of a SPN can be obtained safely with high diagnostic yield. Correlation to detailed clinical data is expected to help selecting patients for this procedure in the future.

In the future add on technique such as confocal laser endomicroscopy and fluorescence molecular endoscopy might further improve identification of the lesion during the procedure. Ultimately, we expect that development of this technique will pave the way to a one-stop-shop approach with rapid on-site evaluation followed by local treatment (e.g. microwave ablation) of the malignant pulmonary nodule.

ELIGIBILITY:
Inclusion Criteria:

* age >18
* pulmonary nodule(s) suspicious for malignancy or metastases of a known primary tumour
* a distinct nodule with a diameter of >6 mm in its largest dimension
* nodule located in the parenchymal tissue >1 cm from the pleura and bronchoscopically accessible through a point of entry
* willing to give informed consent to the procedure.

Exclusion Criteria:

* any contraindication to undergo bronchoscopy
* contraindication for general anaesthesia
* inability to stop anticoagulants or antiplatelets agents according to the UMCG protocol
* childbearing or breastfeeding women
* moderate to seyere pulmonary fibrosis
* severe emphysema with bullae > 5 cm m the vicinity of the target nodule or tunnel.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients undergoing a Virtual bronchoscopy navigation procedure to assess a solitary pulmonary nodule.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Successful diagnostic procedure | During procedure
  Number of procedures with success to access the solitary pulmonary nodule

CONTACTS AND LOCATIONS:
Overall Officials: Dirk-Jan Slebos, MD PhD, Principal Investigator — UMCG Groningen, The Netherlands
Locations (1):
- UMCG Groningen, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided